CLINICAL TRIAL: NCT03319849
Title: A Phase III Multicenter Randomized, Sham Controlled, Study to Determine the Safety and Efficacy of NT-501 in Macular Telangiectasia Type 2
Brief Title: A Study to Determine the Safety and Efficacy of NT-501 in Macular Telangiectasia Type 2 - Protocol B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Collaborators: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTMT-03-B
Record Dates: First submitted 2017-10-03; First posted 2017-10-24 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Macular Telangiectasia Type 2
Keywords: Ciliary Neurotrophic Factor (CNTF); Macular Telangiectasia (MacTel); MacTel
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: After confirming eligibility in conjunction with the reading center, the study eye of each subject was randomized (1:1) to either have NT-501 implanted or to undergo the sham procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects and all personnel at the image reading center remained masked to the treatment assignment throughout the study. In addition, the refractionist, VA examiner, and photographers/imagers were masked to treatment assignment (NT-501 implantation or sham procedure) at all follow-up visits. The ophthalmologist, surgeon, and clinic coordinator were instructed not to discuss the assigned treatment with the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NT-501 (Experimental): Test product
  Interventions: Combination Product: NT-501
- Sham (Sham Comparator): A sham surgical procedure was performed to mimic the implant procedure; there was no comparator product.
  Interventions: Procedure: Sham

INTERVENTIONS:
Combination Product: NT-501 — Each NT-501 implant consisted of hCNTF-secreting NTC-201-6A.02 cells encapsulated within supportive matrices and surrounded by a semipermeable polymer membrane.
  The NTC-201-6A cells continuously secrete CNTF from the NT-501 implant into the vitreous cavity. Implanted by a qualified Health Care Professional.
  Arms: NT-501
Procedure: Sham — The sham surgery involved a superficial conjunctival incision performed under local anesthetic and closure with a single suture.
  Arms: Sham

SUMMARY:
This study is a phase 3, randomized, multi-center study to evaluate the efficacy and safety of the NT-501 implants in participants with macular telangiectasia type 2.

DETAILED DESCRIPTION:
Phase 3, prospective, multicenter, masked, sham-controlled study with the overall study objective to evaluate the efficacy and safety of NT-501 for the treatment of MacTel. Secondary objective was to evaluate the safety of NT-501 in participants with MacTel. This was a multicenter study conducted at 20 study centers in the United States, Australia, Germany, and the United Kingdom.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant must have at least one study eye with a positive diagnosis of MacTel with evidence of fluorescein leakage typical of MacTel and at least one of the other features that include hyperpigmentation that is outside of a 500 micron radius from the center of the fovea, retinal opacification, crystalline deposits, right-angle vessels, or inner/outer lamellar cavities
2. Participant must have an Inner Segment - Outer Segment Junction Line (IS/OS) Photo Receptor (PR) break in the study eye(s) and en face EZ (area of IS/OS loss) as measured by spectral-domain optical coherence tomography (SD-OCT) between 0.16 mm^2 and 2.00 mm^2
3. Participant's best corrected visual acuity (BCVA) is a 54-letter score or better (20/80 or better) as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at screening.
4. Participant must have steady fixation in the foveal or parafoveal area and sufficiently clear media for good quality photographs
5. Participant must be greater than 21 years of age or less than 80 years of age at screening
6. Participant must be able to provide written informed consent to participate in the study, in accordance with the International Conference on Harmonisation Good Clinical Practices guidelines, and local regulations, before initiating any study-related procedures
7. Women of childbearing potential must agree to use highly effective contraception (Germany and France only)

Key Exclusion Criteria:

1. Participant is medically unable to comply with study procedures or follow-up visits
2. Participant received intravitreal steroid therapy for non-neovascular MacTel within the last 3 months
3. Participant has ever received intravitreal anti-vascular endothelial growth factor (VEGF) therapy in the study eye OR has, within the past 3 months, received intravitreal anti-VEGF in the fellow eye at randomization
4. Participant has evidence of ocular disease other than MacTel that, in the judgment of the examining physician, may confound the diagnosis, procedures or outcome of the study (eg, glaucoma, severe nonproliferative or proliferative diabetic retinopathy, uveitis)
5. Participant has a chronic requirement (eg, ≥ 4 weeks at a time) for ocular medications and/or has a diagnosed disease that, in the judgment of the examining physician, may be vision threatening or may affect the primary outcome (artificial tears are permitted)
6. Participant has evidence of intraretinal neovascularization or subretinal neovascularization (SRNV), as evidenced by hemorrhage, hard exudate, subretinal fluid or intraretinal fluid in either eye
7. Participant has evidence of central serous chorio-retinopathy in either eye
8. Participant has evidence of pathologic myopia in either eye
9. Participant has significant corneal or media opacities in either eye
10. Participant has had a vitrectomy, penetrating keratoplasty, trabeculectomy, or trabeculoplasty
11. Participant has any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 2, or a nuclear opacity > standard 3 as measured on the Age-Related Eye Disease Study (AREDS) clinical lens grading system
12. Participant has undergone lens removal in the previous 3 months or YAG laser within 4 weeks
13. Participant was a participant in any other clinical trial of an intervention (drug or device) within the last 6 months
14. Participant is on chemotherapy
15. Participant is pregnant or breastfeeding
16. Participant has a history of malignancy that would compromise the 24-month study survival
17. Participant with a history of ocular herpes virus in either eye
18. Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations, and outcome assessments
19. Participant has evidence of intraretinal hyperreflectivity by OCT

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gillies, MD, Principal Investigator — Save Sight/Sydney, Australia
Locations (27):
- United States (22):
  - Retina Vitreous Assoc, Beverly Hills, California
  - Retina Consultants of Southern Colorado, P.C., Colorado Springs, Colorado
  - Emory University Eye Center, Atlanta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Elman Retina Group, PA, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary Ophthalmology Clinical Research Office, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Retina Institute, Chesterfield, Missouri
  - Retina Center of New Jersey - Envision Ocular, LLC, Bloomfield, New Jersey
  - Flaum Eye - University of Rochester, Rochester, New York
  - University of Rochester Strong Memorial Hospital, Rochester, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Scheie Eye Institute - University of Pennsylvania, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Center of Texas, Southlake, Texas
- Australia (2):
  - Save Sight Institute, Sydney, Sydney, New South Wales
  - Centre for Eye Research Australia Macular Research Unit, East Melbourne, Victoria
- Germany (3):
  - Klinik at Freiberg, Germany, Freiburg im Breisgau, Baden-Wurttemberg Germany
  - University of Bonn, Bonn, North Rhine-Westphalia
  - St. Franziskus, Muenster, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew EY, Gillies M, Jaffe GJ, Gaudric A, Egan C, Constable I, Clemons T, Aaberg T, Manning DC, Hohman TC, Bird A, Friedlander M; MacTel CNTF NTMT-03 Research investigators. Cell-Based Ciliary Neurotrophic Factor Therapy for Macular Telangiectasia Type 2. NEJM Evid. 2025 Aug;4(8):EVIDoa2400481. doi: 10.1056/EVIDoa2400481. Epub 2025 Jul 22. PMID 40693847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening period for up to 30 days
Pre-assignment Details: 119 subjects enrolled (6 participants withdrew after randomization) but prior to the implantation/sham surgery procedure; 59 subjects in NT-501 arm and 54 subjects in sham arm.
Units Other Than Participants: eyes
Groups:
- NT-501: NT-501: Surgery to receive one NT-501 device implant.
- Sham: Sham: Non-penetrating sham procedure to mimic implant procedure.
Period: Overall Study
Arm/Group | NT-501 | Sham
Started | 60; 60 eyes | 59; 59 eyes
Treated (Underwent Surgery) (Participants who actually underwent surgery for either NT-501 or sham treatment) | 59; 59 eyes | 54; 54 eyes
Completed | 57; 57 eyes | 49; 49 eyes
Not Completed | 3; 3 eyes | 10; 10 eyes
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — COVID-19 | 0 | 1
Not completed — Other | 1 | 2
Not completed — Eligible and did not enroll in amendment | 1 | 3
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat population comprised all randomized subjects who underwent surgery (NT-501 implantation or sham surgery) whether or not the subject adhered to the study protocol.
Groups:
- Sham: A sham surgical procedure was performed to mimic the implant procedure; there was no comparator product.
  Sham Procedure: The sham surgery involved a superficial conjunctival incision performed under local anesthetic and closure with a single suture.
- Total: Total of all reporting groups
Arm/Group | NT-501 | Sham | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 36 | 78
  >=65 years | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (7.61) | 58.7 (8.87) | 58.6 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 36 | 82
  Male | 13 | 18 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 55 | 49 | 104
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 47 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Baseline Ocular Characteristics (mITT) - Ocular Visual Acuity [Mean (Standard Deviation); unit: Best-corrected visual acuity (letters)] — Measure Description: BCVA using standard ETDRS
  Best-corrected visual acuity (letters) | 74.4 (7.76) | 73.6 (9.23) | 74.0 (8.47)
Baseline Ocular Characteristics (mITT) - Area of EZ loss (mm^2) [Mean (Standard Deviation); unit: Area of EZ loss (mm^2)] | 0.518 (0.3120) | 0.476 (0.2934) | 0.498 (0.3027)
Baseline Ocular Characteristics (mITT) - Monocular Reading Speed [Mean (Standard Deviation); unit: words per minute] | 96.49 (47.314) | 94.09 (42.806) | 95.36 (45.051)
Baseline Ocular Characteristics (mITT) - Pupil Diameter [Mean (Standard Deviation); unit: Pupil diameter (mm)] | 3.53 (1.130) | 3.90 (1.092) | 3.70 (1.123)
Intraocular Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 15.2 (3.19) | 14.6 (2.70) | 14.9 (2.97)
Natural Lens Present [Count of Participants; unit: Participants]
  Yes | 52 | 46 | 98
  No | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Change in the Area of EZ Area of Loss From Baseline Through Month 24
Description: The rate of change in the area of EZ loss (IS/OS; macular photoreceptor loss) from baseline through month 24, as assessed using SD-OCT in the study eye of participants with MacTel.
Time Frame: End point timeframe is through Month 24. Baseline, Month 6, 12, 16, 20 and 24. Month 6 was collected but not included in the primary analyses.
Population: The efficacy and safety of the NT-501 implant that delivers a daily dose of CNTF in comparison to sham surgery with no implant, in participants with confirmed MacTel.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | NT-501 | Sham
Number analyzed (Participants) | 58 | 57
mm^2 | 0.111 (0.0142) | 0.160 (0.0149)
Statistical Analysis 1: Comparison: NT-501 vs Sham; Test type: Superiority; p = 0.0186, Mixed Models Analysis; Median Difference (Final Values) = -0.049, 95% CI 2-sided [-0.0890 to -0.0082], Standard Error of Mean 0.0206

2. Secondary Outcome: Mean Change in Aggregate Retinal Sensitivity Loss and Aggregate Interpolated Retinal Sensitivity Loss by Microperimetry (mITT Population)
Description: Change from baseline in retinal sensitivity loss as measured by as measured by Macular Integrity Assessment (MAIA)
Time Frame: Baseline through 24 months.
Population: All treated participants (mITT population)
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Aggregate Retinal Sensitivity Loss (dB) - NT-501: Aggregate Retinal Sensitivity Loss (dB) with NT-501 treatment through Month 24
- Aggregate Retinal Sensitivity Loss (dB) - Sham: Aggregate Retinal Sensitivity Loss (dB) with Sham treatment through Month 24
- Aggregate Interpolated Retinal Sensitivity Loss (dB) - NT-501: Aggregate Interpolated Retinal Sensitivity Loss (dB) with NT-501 treatment through Month 24
- Aggregate Interpolated Retinal Sensitivity Loss (dB) - Sham: Aggregate Interpolated Retinal Sensitivity Loss (dB) with sham treatment through Month 24
Arm/Group | Aggregate Retinal Sensitivity Loss (dB) - NT-501 | Aggregate Retinal Sensitivity Loss (dB) - Sham | Aggregate Interpolated Retinal Sensitivity Loss (dB) - NT-501 | Aggregate Interpolated Retinal Sensitivity Loss (dB) - Sham
Number analyzed (Participants) | 59 | 54 | 59 | 54
dB
  Baseline Actual: number analyzed (Participants) | 56 | 53 | 56 | 53
  Baseline Actual | 55.54 (56.050) | 51.84 (57.380) | 34864.17 (35305.260) | 32445.03 (38667.790)
  Month 24 Actual: number analyzed (Participants) | 52 | 48 | 52 | 48
  Month 24 Actual | 97.77 (78.620) | 93.02 (70.414) | 61076.49 (52619.379) | 58360.26 (50535.070)
  Month 24 Change from Baseline: number analyzed (Participants) | 52 | 48 | 52 | 48
  Month 24 Change from Baseline | 40.02 (51.278) | 41.97 (41.111) | 24859.88 (31165.862) | 26309.32 (25374.040)

3. Secondary Outcome: Monocular Reading Speed (mITT Population)
Description: Change from baseline through Month 24 for Monocular reading speed assessed using International Reading Speed Texts (IReST) cards developed by the IReST Study Group 21
Time Frame: Baseline through 24 months.
Population: All treated participants (mITT population) without missing data
Measure: Mean (Standard Deviation); unit: Reading Speed (words per minute)
Arm/Group | NT-501 | Sham
Number analyzed (Participants) | 59 | 54
Reading Speed (words per minute)
  Baseline Actual | 96.49 (47.314) | 94.09 (42.806)
  Month 24 Actual | 92.18 (45.090) | 77.33 (43.899)
  Month 24 Change from Baseline | -5.46 (29.648) | -18.88 (33.705)

ADVERSE EVENTS:
Time Frame: During the Clinical Trial
Description: Any non-ocular events and/or ocular events in the study eye.
Arm/Group | NT-501 | Sham
All-Cause Mortality (participants affected / at risk) | 1/59 | 0/54
Serious Adverse Events (participants affected / at risk) | 11/59 | 10/54
Other Adverse Events (participants affected / at risk) | 56/59 | 48/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NT-501 (N=59) | Sham (N=54)
Suture related complication (Injury, poisoning and procedural complications) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Device extrusion (Product Issues) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NT-501 (N=59) | Sham (N=54)
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypertension (Vascular disorders) | 4 | 1
Hot flush (Vascular disorders) | 0 | 2
Prehypertension (Vascular disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Adverse drug reaction (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Menopause (Social circumstances) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Product deposit (Product Issues) | 1 | 0
Intraocular pressure increased (Investigations) | 2 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Mammogram abnormal (Investigations) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 14 | 2
Conjunctival scar (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Macular dystrophy congenital (Congenital, familial and genetic disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Aura (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Ageusia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 19 | 10
Foreign body sensation in eyes (Eye disorders) | 14 | 8
Conjunctival hyperaemia (Eye disorders) | 12 | 7
Eye pain (Eye disorders) | 12 | 6
Delayed dark adaptation (Eye disorders) | 15 | 2
Conjunctival oedema (Eye disorders) | 4 | 6
Vision blurred (Eye disorders) | 6 | 3
Dry eye (Eye disorders) | 6 | 2
Miosis (Eye disorders) | 8 | 0
Conjunctival irritation (Eye disorders) | 3 | 3
Swelling of eyelid (Eye disorders) | 3 | 3
Visual impairment (Eye disorders) | 3 | 3
Vitreous floaters (Eye disorders) | 6 | 0
Vitreous haemorrhage (Eye disorders) | 6 | 0
Choroidal neovascularisation (Eye disorders) | 2 | 1
Eye irritation (Eye disorders) | 2 | 3
Metamorphopsia (Eye disorders) | 1 | 4
Ocular discomfort (Eye disorders) | 4 | 1
Eye discharge (Eye disorders) | 2 | 1
Eye pruritus (Eye disorders) | 2 | 1
Lacrimation increased (Eye disorders) | 0 | 3
Retinal haemorrhage (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 2 | 0
Anterior chamber cell (Eye disorders) | 2 | 0
Anterior chamber flare (Eye disorders) | 2 | 0
Asthenopia (Eye disorders) | 0 | 2
Blepharitis (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Cataract subcapsular (Eye disorders) | 2 | 0
Diplopia (Eye disorders) | 2 | 0
Meibomian gland dysfunction (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 0 | 2
Photopsia (Eye disorders) | 1 | 1
Punctate keratitis (Eye disorders) | 1 | 1
Visual field defect (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Anterior chamber collapse (Eye disorders) | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1
Cataract cortical (Eye disorders) | 1 | 0
Chorioretinal folds (Eye disorders) | 1 | 0
Conjunctival cyst (Eye disorders) | 1 | 0
Corneal deposits (Eye disorders) | 1 | 0
Corneal epithelium defect (Eye disorders) | 1 | 0
Corneal erosion (Eye disorders) | 0 | 1
Corneal opacity (Eye disorders) | 0 | 1
Delayed light adaptation (Eye disorders) | 1 | 0
Epiretinal membrane (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 1 | 0
Eyelid margin crusting (Eye disorders) | 1 | 0
Eyelid pain (Eye disorders) | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 1
Hypotony of eye (Eye disorders) | 1 | 0
Lenticular opacities (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Night blindness (Eye disorders) | 0 | 1
Periorbital pain (Eye disorders) | 1 | 0
Pinguecula (Eye disorders) | 1 | 0
Presbyopia (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 1 | 0
Retinal vasculitis (Eye disorders) | 1 | 0
Scleral thinning (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Vitreoretinal traction syndrome (Eye disorders) | 1 | 0
Vitreous haze (Eye disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Periodontal inflammation (Gastrointestinal disorders) | 1 | 0
Tooth erosion (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3
COVID-19 (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 2
Ear infection (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Candida infection (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pilonidal disease (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site agrees not to make any publication prior to Sponsor's initial publication. Site agrees that proposed manuscripts, abstracts, or oral presentations relating to the Study Drug will be submitted directly to Sponsor at least sixty (60) days prior to submission for publication or presentation to ensure that Confidential Information (including Clinical Data or Study results not disclosed in Sponsor's prior publication), Sponsor Technology or Sponsor-Owned Inventions are protected.

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT03319849/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03319849/SAP_001.pdf